CLINICAL TRIAL: NCT03637699
Title: A Phase I Randomized Controlled Trial of a Positive Psychology Intervention for Patients With Multiple Sclerosis
Brief Title: A Positive Psychology Intervention for Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Consortium of Multiple Sclerosis Centers (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Bonnie Ilene Glanz, Research Associate, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P002375
Record Dates: First submitted 2018-08-06; First posted 2018-08-20 (Actual); Results first posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: Positive Psychology; Positive Affect
MeSH Terms: conditions — Multiple Sclerosis | interventions — Psychology, Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Subjects randomized to the intervention group will be complete five weeks of positive psychology exercises, one exercise per week, during the intervention phase (weeks 1-5) of the study.
  Interventions: Behavioral: Positive Psychology
- Waitlist Control (Other): Subjects randomized to the waitlist control group will complete five weeks of positive psychology exercises, one exercise per week, during the extension phase (weeks 6-10) of the study.
  Interventions: Behavioral: Positive Psychology

INTERVENTIONS:
Behavioral: Positive Psychology — 5-week positive psychology intervention

SUMMARY:
Positive psychology (PP) uses targeted activities to increase the frequency and intensity of positive emotional experiences such as positive affect. Examples of PP activities include recalling positive life events and performing acts of kindness. This pilot study will examine the tolerability and efficacy of a PP training program to increase positive affect in patients with multiple sclerosis (MS). In the intervention phase, subjects randomized to the intervention group will complete five weeks of PP exercises, one exercise per week. Subjects will also have weekly calls with the study trainer. The control group will have no study activities. In the extension phase, subjects in the control group will complete PP training as described above. The investigators will examine the tolerability of the program by calculating the proportion of subjects who complete the program. The investigators will also examine exercise-specific ratings of ease and utility to measure the acceptability of each exercise. Finally, the investigators will evaluate the efficacy of PP training by comparing subjects in the intervention and control groups on measures of positive affect, emotional function, health-related quality of life (HRQOL) and self-reported functional activities such as work. If successful, this study will advance the use of PP as a low cost, innovative and effective tool for increasing positive affect, decreasing depression and anxiety and improving HRQOL in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis according to the McDonald 2010 diagnostic criteria
* Age 18-65
* Ability to speak, read and write in English
* Enrollment in the Comprehensive Longitudinal Investigation of Multiple Sclerosis at the Brigham and Women's Hospital, Partners MS Center: The CLIMB Study.

Exclusion Criteria:

• Moderate or marked cognitive abnormalities on brief mental status testing identified that would preclude meaningful participation in the PP exercises.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Waitlist Control
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Subjects randomized to the intervention group will complete five weeks of positive psychology exercises, one exercise per week, during the intervention phase (weeks 1-5) of the study.
  Positive Psychology: 5-week positive psychology intervention
- Total: Total of all reporting groups
Arm/Group | Intervention | Waitlist Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (7.2) | 54.2 (4.7) | 54.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of PP Exercises Completed by Subjects
Description: Measured by percentage of PP exercises completed by subjects.
Time Frame: Five weeks
Measure: Number; unit: percentage of exercises completed
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 15 | 15
percentage of exercises completed | 93 | 93

2. Secondary Outcome: Subject Ratings of Ease of Completion of PP Exercises
Description: Measured by weekly 0-10 post-exercise Likert scale ratings of ease of completion of PP exercise provided by subjects, with 0 being very difficult to complete and 10 being very easy to complete. Scores range from 0-10.
Time Frame: Five weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Gratitude for positive events | 9.0 (1.3) | 8.4 (1.9)
  Personal strengths | 8.1 (2.2) | 7.5 (2.2)
  Gratitude letter | 7.8 (1.8) | 7.6 (2.1)
  Enjoyable and meaningful activities | 9.1 (1.5) | 8.2 (1.7)
  Remembering past successes | 8.4 (1.3) | 9.0 (1.1)

3. Secondary Outcome: Changes in Affect
Description: Measured by the Positive and Negative Affect Schedule (PANAS). PANAS is comprised of two 10-item mood scales, one measuring positive affect and the other measuring negative affect. Scores on the Positive Affect scale range from 10-50. Higher scores are associated with greater positive affect. Scores on the Negative Affect scale range from 10-50, with lower scores representing lower levels of negative affect.
Time Frame: Five weeks
Population: Missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Positive affect: number analyzed (Participants) | 12 | 13
  Positive affect | 4.9 (4.5) | -3.2 (5.8)
  Negative affect: number analyzed (Participants) | 13 | 11
  Negative affect | -2.6 (9.4) | -0.3 (4.5)

4. Secondary Outcome: Change in Trait Optimism
Description: Measured by the Life Orientation Test - Revised (LOT-R). LOT-R is a 6-item measure of trait optimism and pessimism. Scores range from 0-24. Higher scores are associated with greater optimism.
Time Frame: Five weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 14 | 14
score on a scale | 2.1 (3.4) | -1.3 (2.5)

5. Secondary Outcome: Change in Depression
Description: Measured by the Center for Epidemiologic Studies Depression Scale (CES-D). CES-D is a 20-item measure of depression with scores ranging from 20-80. Higher scores are associated with greater depression.
Time Frame: Five weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 14 | 12
score on a scale | -2.1 (2.9) | 0 (5.7)

6. Secondary Outcome: Change in Anxiety
Description: Measured by the State Trait Anxiety Inventory (STAI). STAI includes two 20-item questionnaires designed to measure the current temporary condition of "state" anxiety and the more general and longstanding condition of "trait" anxiety. Scores for each scale range from 20-80. Higher scores are associated with greater anxiety.
Time Frame: Five weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 14 | 14
score on a scale
  State anxiety | -3.2 (6.1) | 3.4 (8.1)
  Trait anxiety | -3.3 (4.9) | 2.7 (6.9)

7. Secondary Outcome: Changes in Health-related Quality of Life
Description: Measured by the Medical Outcomes Study Short Form (SF-36). The SF-36 is a 36-item measure of health status and quality of Life. It consists of eight scaled scores and two summary scores. The lower the score, the more disability. The higher the score, the less disability. Scores for each scale range from 0-100.
Time Frame: Five weeks
Population: Missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Physical functioning: number analyzed (Participants) | 11 | 13
  Physical functioning | -1.0 (3.3) | 0.3 (3.2)
  Role physical: number analyzed (Participants) | 14 | 13
  Role physical | 4.2 (6.3) | 1.1 (9.0)
  Bodily pain | 0.1 (8.3) | -0.2 (7.5)
  General health | 1.1 (4.0) | -2.9 (3.9)
  Vitality | 1.4 (4.2) | 0.3 (7.7)
  Social functioning: number analyzed (Participants) | 13 | 14
  Social functioning | 3.0 (6.7) | 2.4 (9.2)
  Role emotional | -3.6 (9.4) | -4.3 (12.3)
  Mental health | 2.9 (4.6) | -0.8 (6.6)
  Physical component summary: number analyzed (Participants) | 11 | 13
  Physical component summary | 0.9 (4.2) | 0.3 (5.4)
  Mental component summary: number analyzed (Participants) | 11 | 13
  Mental component summary | 0.5 (6.0) | -1.4 (6.3)

8. Secondary Outcome: Change in Work Productivity
Description: Measured by the Work Productivity and Activity Impairment Questionnaire (WPAI). Outcomes are expressed as impairment percentages with higher scores indicating greater impairment and less productivity. Scores range from 0-100.
Time Frame: Five weeks
Population: Work time missed, Work impairment and Overall work impairment are only completed by subjects who are employed. Missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 14 | 14
score on a scale
  Work time missed: number analyzed (Participants) | 9 | 6
  Work time missed | -1.0 (4.9) | -1.9 (10.8)
  Work impairment: number analyzed (Participants) | 8 | 6
  Work impairment | 1.2 (24.7) | 3.3 (10.3)
  Overall work impairment: number analyzed (Participants) | 9 | 6
  Overall work impairment | 0.1 (22.1) | 0.5 (15.6)
  Activity impairment | 0 (26.9) | 5.0 (23.5)

9. Secondary Outcome: Change in Perceived Stress
Description: Measured by the Perceived Stress Scale (PSS). The PSS is a 10-item questionnaire with scores ranging from 0-40. Higher scores are associated with greater perceived stress.
Time Frame: Five weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 14 | 14
units on a scale | -0.4 (2.8) | -1.1 (2.7)

10. Secondary Outcome: Change in Resilience
Description: Measured by the Brief Resilience Scale (BRS). The BRS is a 6-item measure of resilience with scores ranging from 1-5. Higher scores are associated with greater resilience.
Time Frame: Five weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 13 | 14
score on a scale | 0.1 (0.4) | -0.3 (0.5)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Intervention | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
This study had a small sample size and a large number of outcome measures which may limit the ability to see statistically significant changes in health-related quality of life and other psychological outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT03637699/Prot_SAP_000.pdf